CLINICAL TRIAL: NCT00180570
Title: Scandinavian Atrial Lead Trial
Brief Title: SALT - Success of Active Versus Passive Lead Fixation of Atrial Pacing/Sensing Electrodes
Acronym: SALT
Status: Suspended | Phase: Phase 4 | Type: Interventional
Sponsor: Guidant Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SALT-2
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2005-09

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

INTERVENTIONS:
Device: FineLine II Sterox, FineLine II Sterox, FineLine II Sterox EZ

SUMMARY:
Randomised Comparison with regards to complication rate and electrical measurements of atrial leads with different fixation mechnism

DETAILED DESCRIPTION:
This investigation will study and compare 3 types of electrically identical, commercially available FineLine II Sterox leads with different fixation mechanisms. This trial has been designed to primarily study the difference in repositioning rate between active and passive fixation (straight and J-shaped) leads, if any. It will also monitor and document the behavior of the study leads, with special reference to electrical parameters and handling. Normal measurements are taken at pre-dicharge, 1-month 3-month and 12-month follow-up

ELIGIBILITY:
Inclusion Criteria:

* Patients selected for participation in this investigation should be candidates for permanent pacemaker implantation chosen from the investigator's general patient population without regard for race or sex. Furthermore, these patients should, in the physician's general opinion, benefit from permanent pacemaker implantation with one of the study leads. Patients should be geographically stable and available for routine follow-up visits throughout the duration of the study. Patients must also be able and willing to provide informed consent.

Exclusion Criteria:

* Patients who previously went through heart surgery should be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385
Dates: Start 1997-01; Study Completion 2006-01

PRIMARY OUTCOMES:
The primary objective of this study is to compare repositioning rate due to threshold > 3.0 V @ 0.5 ms or P-wave < 0.8 mV between FineLine II Sterox 4480 and 4470, and between 4456 and 4470.

SECONDARY OUTCOMES:
1. Other complications (Safety). To compare other lead related complication rates such as perforation, lead fracture and failure to implant. 2. Electrical properties

CONTACTS AND LOCATIONS:
Overall Officials: charles kennergren, Principal Investigator — Sahlgrenska Sjukhuset i Göteborg Sweden
Locations (1):
- Sahlgrenska Sjukhuset i Göteborg Sweden,, Gothenburg, Sweden